CLINICAL TRIAL: NCT05631314
Title: Lets Agree to Disagree on Operative Versus Nonoperative (LADON) Treatment for Distal Radius Fractures in the Elderly - a Prospective International Multicenter Cohort Study
Brief Title: Lets Agree to Disagree on Operative vs Nonoperative Treatment for Distal Radius Fractures in the Elderly (LADON Radius)
Acronym: LADON radius
Status: Not yet recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Arthrex GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: LADON radius
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Radius Fracture Distal
Keywords: distal radius fracture; elderly; operative treatment; natural experiment
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operative treatment: This group will consist of patients who underwent operative treatment for a distal radius fracture.
  Interventions: Procedure: operative treatment
- non-operative treatment: This group will consist of patients who underwent non-operative treatment for a distal radius fracture.
  Interventions: Procedure: non-operative treatment

INTERVENTIONS:
Procedure: operative treatment — Operative treatment can consist of open reduction and volar and/or dorsal plating or closed reduction and fixation with K-wires, external fixateur.
  Groups: operative treatment
Procedure: non-operative treatment — Non-operative treatment will consist of immobilization in a below the elbow cast for 4-6 weeks with or without prior closed reduction.
  Groups: non-operative treatment

SUMMARY:
The primary objective of this study is to determine if non-operative treatment of distal radius fractures in patients aged 65 and over leads to equal funtional results as operative treatment. To do so patients will be included from two "schools" in which treatment i seither predominantly operative or non-operative. There will be no study intervention as patients will be treated as per local standard of care. The study is set up as an international multicenter study. Those patients included in the study will be follow-up at 6 weeks, 12 weeks, 1 year and 2 years after treatment was initiated. Our hypothesis is, that patients treated operatively will have better function than those treated non-operatively.

DETAILED DESCRIPTION:
This study is an international multicenter prospective observational cohort study for which patients will be identified after treatment has been initiated. Outcome data will be prospectively collected. Patients will be recruited from five hospitals in countries with a predominant preference for operative (Switzerland, "School" A) and non-operative treatment (the Netherlands, "School" B). After a treatment plan has been established, patients will be approached either during the index hospital admission or during one of their follow-up appointments in the outpatient clinic within six weeks to explain the purpose and procedures of the study. Patients will be asked to provide written informed consent. Following the identification of eligible patients, anonymous radiographs including key images of CT-scans if available and baseline characteristics (such as age, co-morbidities, activity level) as well as relevant laboratory results will be made available to the expert panel (details below) on a secure online platform. This will allow the members of the panel to reach a "clinical" decision regarding their treatment recommendation. The panel will be blinded to the actual treatment received and the origin of the case.

The expert panel will consist of three representatives from both "Schools". All panel members will be certified trauma surgeons from one of the participating hospitals. Eligible patients will be reviewed by the experts every two weeks. Patients will ultimately be included in the study if clinical equipoise is achieved, meaning the majority of experts in one "School", minimally two out of three, disagree with the received treatment in the other "School". For example, eligible patients would have received operative treatment based on the expert opinions in "School" A, however, were in fact treated non-operatively according to the treating surgeon in "School" B and vice versa. If the majority of the panel in one "School" agree with the received treatment in the other "School" the patient will be excluded. This will lead to two comparable groups for which true clinical equipoise exists. The actual treatment the patient receives, will continue as initially planned by the treating hospital.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* acute (< 14 days after injury) distal radius fracture
* treated at one of the participating hospitals

Exclusion Criteria:

* initial operative treatment at a non-participating hospital
* delayed presentation (>14 days after injury)
* patient actively refuses the recommended treatment
* insufficient follow-up (<12 months) or unavailable to follow-up due to residency in other hospital area
* concomitant injury to the ipsilateral or contralateral upper extremity
* cognitive impairment precluding answering questionnaires
* non-German, non-English, non-Dutch speaking
* pre-existing co-morbidities which preclude operative treatment
* pathological fractures
* open fractures
* neurovascular injury requiring operative treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients presenting to the emergency department or out-patient clinic in one of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
PRWE 12 weeks | 12 weeks
  Patient-rated Wrist Evaluation scores measured a t 12 weeks after treatment initiation

SECONDARY OUTCOMES:
PRWE 1 and 2 years | 1 year, 2 years
  Patient-rated Wrist Evaluation scores measured 1 and 2 years after treatment initiation
PASE | 12 weeks, 1 year, 2 years
  Physical activity score of the elderly
Pain intensity | 6 weeks, 12 weeks, 1 year, 2 years
  numeric rating system for pain
range of motion | 12 weeks, 1 year, 2 years
  range of motion of the wrist
EQ-5D-5L | 12 weeks, 1 year, 2 years
  Quality of life score
Complications | 6 weeks, 12 weeks, 1 year, 2 years
  Complications will be assessed. They will include infection, non-union, implant failure, complex regional pain syndrome and any adverse event need surgical intervention. For patients treated surgically, the need for implant removal will also be recorded.
living situation | 6 weeks, 12 weeks, 1 year, 2 years
  the living situation of the patient will be assessed and classified as one of the following categories: independent, independent with support from family/district nurse or similar, nursing home.
radiological outcome | 6 weeks, 12 weeks, 1 year, 2 years
  The xrays will be assessed to judge the radiological outcome with regards to loss of reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Frank JP Beeres, PD PhD, Principal Investigator — Luzerner Kantonsspital